CLINICAL TRIAL: NCT03972774
Title: Assessment of Patients With suspeCted Coronary Artery Disease by Coronary calciUm fiRst strATegy vErsus Usual Care Approach
Acronym: ACCURATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1051080
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac PET stress testing and test-dependent management (Other): Subjects randomized to the cardiac PET stress test strategy will receive appropriate subsequent care depending on the outcome of the cardiac PET scan (i.e., depending on whether ischemia is present or not).
  Interventions: Diagnostic Test: PET Stress Test
- Management without stress-imaging (Other): Subjects randomized to the CAC-only arm will receive appropriate non-PET driven medical clinical management and follow-up.
  Interventions: Other: Non-PET Medical Management

INTERVENTIONS:
Diagnostic Test: PET Stress Test — Cardiac positron emission tomography (PET)/computed tomography (CT) and test-result dependent management
  Arms: Cardiac PET stress testing and test-dependent management
Other: Non-PET Medical Management — Appropriate medical management without cardiac PET stress-imaging
  Arms: Management without stress-imaging

SUMMARY:
The cost of medical care in the United States far exceeds that of all other advanced economies and continues to accelerate at a rate unacceptable to our society, due primarily to the high costs of new imaging technologies and novel drugs (1). Cardiac positron emission tomography (PET) imaging is a powerful new modality for the non-invasive detection of provocable coronary ischemia in patients with low to intermediate-risk chest pain or its equivalent. Intermountain Medical Center (IMC) is performing approximately 6000 clinical cardiac PET scans annually. However, cardiac PET scans are expensive (i.e., billed at >$5,000/scan, average receivable revenue $1500-$2000/scan). Coronary artery calcium (CAC) is a sensitive marker of coronary atherosclerosis. A CAC scan (CACS), performed by multislice computed tomography (CT), is a relatively inexpensive (~$70-$150/scan), low-radiation dose test that marks the presence of coronary atherosclerotic plaque. The absence of CAC has been shown to be associated with very low coronary risk. ACCURATE will test whether a CAC-first strategy (i.e., risk stratification, when CAC ≤ 1, to medical management or to cardiac PET stress testing), performed routinely in symptomatic patients presenting for evaluation of possible coronary artery disease (CAD) prior to the cardiac PET stress test, can be used as a gatekeeper for progression to the expensive rubidium-PET stress (regadenoson) perfusion scan and be a major cost-saver without adversely affecting patient care or outcomes. Routinely, qualifying patients undergo CACS when they present for evaluation of possible but unknown CAD status and are referred for cardiac PET stress testing. In ACCURATE, those with CACS≤1 will then be consented and randomized to either a cardiac PET stress test strategy or a non-PET-driven medical care strategy. Subjects randomized to the cardiac PET stress test strategy will receive appropriate subsequent care depending on the outcome of the cardiac PET scan (i.e., depending on whether ischemia is present or not). Subjects randomized to the CAC-only arm will receive appropriate non-PET driven medical clinical management and follow-up. All participating subjects' electronic medical records will be reviewed indefinitely for clinical outcomes. Initial outcomes will be reported at 1-year, 2-years, and 5-years, with future analyses to be determined by the study investigators.

The objective of this study is to test the hypothesis that PET stress test strategy will results in a decreasing in major adverse cardiac endpoint without exceeding $100,000 per quality-adjusted life year compared to a CAC-first strategy for screening suspected/possible coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥50 years old (i.e., to be of sufficiently high pre-test coronary risk)
* Cardiac PET regadenoson stress perfusion test has been ordered to assess a possible ischemic etiology of low/intermediate risk chest pain or equivalent symptoms (e.g., exertional dyspnea).
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures
* CAC score of ≥1 per routine CAC first strategy (described above)

Exclusion Criteria:

1. Disease history: If available for any of the following diseases: prior known CAD, heart transplant, LVAD, untreated severe valve disease (i.e., severe mitral stenosis, severe mitral regurgitation, and/or severe aortic stenosis), or decompensated heart failure (DHF).
2. Those with a prior CAC score >1.
3. CAC ≤1 prior to this current episode of cardiac assessment

   * Who ELECT to not receive an updated CAC evaluation OR their referring clinician specifically prefers cardiac PET.
   * CAC evaluation repeated at this current episode of cardiac assessment and is now >1.
4. Evidence of possible acute coronary syndrome based on an elevated troponin I ≥0.04ng/mL and/or acute ECG changes of ischemia.
5. Life expectancy <1 year, as assessed by the investigator(s)
6. Cardiac PET/CT is ordered in the pre-operative risk assessment in higher risk non-thoracic surgery.
7. Cardiac PET/CT is ordered for assessment of underlying ischemia in those with arrhythmia to guide anti-arrhythmic therapy.
8. Other conditions that in the opinion of the study investigators and/or referring clinician may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Non-inferior major adverse cardiac endpoint (MACE) outcomes | 1 year
  Routine cardiac PET stress test strategy will result in significantly fewer major adverse cardiac endpoint (MACE) outcomes (defined as coronary death, non-fatal myocardial infarction, cardiac arrest, or ischemia driven revascularization) at 1 year compared with a a CAC-first strategy.
Cost-effectiveness | 5 years
  The costs of routine cardiac PET stress test strategy will be less than <$100,000 per quality-adjusted life year (QALY) compared to CAC-first strategy. Cost-effectiveness, categorized by the American Heart Association, will be defined as achieving at least fair cost effectiveness, i.e., as achieving <$100,000/QALY, which is widely accepted as a "willingness-to-pay" threshold, with <$50,000/QALY defined as good cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk U Knowlton, MD, Principal Investigator — Intermountain Medical Center; Jeffrey L Anderson, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Healthcare Hospitals and Clinics, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided